CLINICAL TRIAL: NCT03016325
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Dose-Ranging, Phase 2b Study of the Safety and Efficacy of Continuous 48-Hour Intravenous Infusions of BMS-986231 in Hospitalized Patients With Heart Failure and Impaired Systolic Function
Brief Title: Evaluate the Safety and Efficacy of 48-Hour Infusions of HNO (Nitroxyl) Donor in Hospitalized Patients With Heart Failure
Acronym: STANDUP AHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV013-011; 2016-001685-29 (EudraCT Number)
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Cohort 1 HNO Donor (Experimental)
  Interventions: Drug: HNO Donor
- Placebo Part 1 Cohort 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2 Cohort 2 HNO Donor- low dose (Experimental)
  Interventions: Drug: HNO Donor
- Part 2 Cohort 2 HNO Donor- high dose (Experimental)
  Interventions: Drug: HNO Donor
- Placebo Part 2 Cohort 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HNO Donor — Infusion
  Other Names: BMS-986231
  Arms: Part 1 Cohort 1 HNO Donor; Part 2 Cohort 2 HNO Donor- high dose; Part 2 Cohort 2 HNO Donor- low dose
Drug: Placebo — Infusion
  Arms: Placebo Part 1 Cohort 1; Placebo Part 2 Cohort 2

SUMMARY:
A Study to Evaluate Safety and Efficacy of Continuous 48-Hour Intravenous Infusions of HNO Donor in Hospitalized Patients with Heart Failure and Impaired Systolic Function

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Actively being hospitalized for acute decompensated heart failure
* At least 1 administration of IV diuretic for the current episode
* Be randomized within 18 hours of first dose of IV diuretic for current episode for Part 1 Cohort 1, or 48 hours for first dose for Part II Cohort II
* Have shortness of breath at rest or with minimal exertion after administration of 1 dose of IV diuretic
* Have history of heart failure and a left ventricular ejection fraction (LVEF) ≤ 40%

Exclusion Criteria:

* Systolic blood pressure <105mm Hg or >160mm Hg or heart rate <50 or >130 bpm
* Have an active infection requiring IV anti-microbial treatment
* Be hospitalized with acute coronary syndrome, coronary revascularization or acute myocardial infarction during the previous 90 days prior to screening
* Have a history of a cerebral vascular accident (CVA or stroke) or of a transient ischemic attack (TIA) during the previous 90 days prior to screening
* Suspected acute lung disease (e.g pneumonia or asthma) or severe chronic lung disease (e.g. severe chronic obstructive pulmonary disease, or pulmonary fibrosis)

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (99):
- United States (24):
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - DMC Detroit Receiving Hospital, Detroit, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Wexner Medical Center at The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Ben Taub General Hospital, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
- Argentina (6):
  - Local Institution, CABA, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Buenos Aires
  - Local Institution, Corrientes
  - Local Institution, Córdoba
  - Local Institution, Santa Fe
- Canada (3):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Québec, Quebec
- Czechia (5):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Plzen-Bory
  - Local Institution, Prague
  - Local Institution, Slaný
- France (7):
  - Local Institution, Besançon
  - Local Institution, Béziers
  - Local Institution, Bobigny
  - Local Institution, Créteil
  - Local Institution, Évreux
  - Local Institution, La Tronche
  - Local Institution, Paris
- Germany (10):
  - Local Institution, Bad Nauheim
  - Local Institution, Frankfurt
  - Local Institution, Göttingen
  - Local Institution, Greifswald
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Homburg
  - Local Institution, Ludwigshafen
  - Local Institution, Mainz
  - Local Institution, Regensburg
- Greece (6):
  - Local Institution, Athens
  - Local Institution, Athens, Attiki
  - Local Institution, Ioannina
  - Local Institution, Kallithea
  - Local Institution, Larissa
  - Local Institution, Thessaloniki
- Italy (3):
  - Local Institution, Brescia
  - Local Institution, Ferrara
  - Local Institution, Foggia
- Japan (14):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Seto, Aichi-ken
  - Local Institution, Fukushima, Fukushima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Amagasaki, Hyōgo
  - Local Institution, Sagamihara-shi, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Suita-shi, Osaka
  - Local Institution, Kawaguchi, Saitama
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Itabashi-ku, Tokyo
  - Local Institution, Osaka
  - Local Institution, Tokyo
- Netherlands (4):
  - Local Institution, Amersfoort
  - Local Institution, Deventer
  - Local Institution, Hardenberg
  - Local Institution, Leeuwarden
- Poland (7):
  - Local Institution, Bialystok
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
  - Local Institution, Zamość
- Spain (6):
  - Local Institution, Alicante
  - Local Institution, Barcelona
  - Local Institution, L'Hospitalet de Llobregat
  - Local Institution, Madrid
  - Local Institution, Sant Joan Despí
  - Local Institution, Santiago de Compostela
- United Kingdom (4):
  - Local Institution, Belfast
  - Local Institution, Blackpool
  - Local Institution, Glasgow
  - Local Institution, London

REFERENCES:
- [Derived] Felker GM, McMurray JJV, Cleland JG, O'Connor CM, Teerlink JR, Voors AA, Belohlavek J, Bohm M, Borentain M, Bueno H, Cole RT, DeSouza MM, Ezekowitz JA, Filippatos G, Lang NN, Kessler PD, Martinez FA, Mebazaa A, Metra M, Mosterd A, Pang PS, Ponikowski P, Sato N, Seiffert D, Ye J. Effects of a Novel Nitroxyl Donor in Acute Heart Failure: The STAND-UP AHF Study. JACC Heart Fail. 2021 Feb;9(2):146-157. doi: 10.1016/j.jchf.2020.10.012. Epub 2020 Nov 25. PMID 33248986
- [Derived] Cowart D, Venuti RP, Lynch K, Guptill JT, Noveck RJ, Foo SY. A Phase 1 Randomized Study of Single Intravenous Infusions of the Novel Nitroxyl Donor BMS-986231 in Healthy Volunteers. J Clin Pharmacol. 2019 May;59(5):717-730. doi: 10.1002/jcph.1364. Epub 2019 Jan 31. PMID 30703258
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Main study cohorts: 100 participants in Part I and 222 in Part II were assigned to treatment (322 randomized in total), of which 97 and 214, respectively, were treated (311 total treated). Reasons not treated (Part I): 3 other reasons. Reasons not treated (Part II): 2 no longer met study criteria; 1 adverse event (AE); 5 other reasons.
  Japanese-specific cohort: 18 participants were randomized and treated in Part II (Japan cohort)
Groups:
- Placebo - Part I: Escalating dose of placebo (3 µg/kg/min for 4 hours, then 6 µg/kg/min for another 4 hours, then 12 µg/kg/min for the remaining 40 hours)
- BMS-986231 - Part I: Escalating dose of BMS-986231 (3 µg/kg/min for 4 hours, then 6 µg/kg/min for another 4 hours, then 12 µg/kg/min for the remaining 40 hours)
- Placebo - Part II: Matching placebo dose of 6 µg/kg/min or 12 µg/kg/min for 48 hours
- BMS-986231 6 µg/kg/Min - Part II: BMS-986231 dose of 6 µg/kg/min for 48 hours
- BMS-986231 12 µg/kg/Min - Part II: BMS-986231 dose of 12 µg/kg/min for 48 hours
- Placebo - Part II (Japan Cohort): Matching placebo dose of 6 µg/kg/min or 12 µg/kg/min for 48 hours for Japanese participants
- BMS-986231 6 µg/kg/Min - Part II (Japan Cohort): BMS-986231 dose of 6 µg/kg/min for 48 hours for Japanese participants
- BMS-986231 12 µg/kg/Min - Part II (Japan Cohort): BMS-986231 dose of 12 µg/kg/min for 48 hours for Japanese participants
Period: Treatment Period
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Started (Started = Entering treatment period) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Completed (Completed = Finished 120 hour treatment period) | 48 | 48 | 70 | 71 | 70 | 6 | 6 | 6
Not Completed | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Participant refuses assessments | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: 32-Day Follow-Up Period
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Started (Started = Entering treatment period) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Completed (Completed = Finished 32-day follow-up period) | 44 | 47 | 62 | 63 | 64 | 6 | 5 | 6
Not Completed | 4 | 2 | 9 | 8 | 8 | 0 | 1 | 0
Not completed — Death | 2 | 0 | 5 | 6 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Poor/non-compliance | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Participant refused to visit | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Family doctor OK'd participant, per call | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — withdrew from Day 5, D32 form not done | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: 182-Day Follow-Up Period
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Started (Started = Entering treatment period) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Completed (Completed = Finished 182-day follow-up period) | 44 | 45 | 60 | 58 | 60 | 1 | 2 | 1
Not Completed | 4 | 4 | 11 | 13 | 12 | 5 | 4 | 5
Not completed — Death | 3 | 3 | 11 | 12 | 9 | 0 | 0 | 1
Not completed — Alive, per national insurance system | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Alive, per Family doctor | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Alive, per civil unit | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Vital status collected via EMR | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — withdrew from D5, D32/182 forms not done | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No cont D182 FU, Sponsor admin reason | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort) | Total
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6 | 329
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (12.23) | 64.6 (12.23) | 67.3 (11.52) | 69.2 (11.41) | 70.0 (11.52) | 65.3 (17.88) | 69.5 (13.31) | 76.7 (10.48) | 67.9 (11.94)
Age, Customized [Count of Participants; unit: Participants] — Age categorical
  Participants
    < 65 years | 17 | 24 | 21 | 23 | 19 | 3 | 3 | 1 | 111
    65 -to <=75 years | 22 | 15 | 36 | 26 | 30 | 0 | 1 | 2 | 132
    >75 years | 9 | 10 | 14 | 22 | 23 | 3 | 2 | 3 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18 | 20 | 15 | 0 | 1 | 2 | 74
  Male | 40 | 39 | 53 | 51 | 57 | 6 | 5 | 4 | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 9 | 11 | 11 | 0 | 0 | 0 | 32
  Not Hispanic or Latino | 44 | 45 | 18 | 23 | 20 | 0 | 0 | 0 | 150
  Unknown or Not Reported | 4 | 3 | 44 | 37 | 41 | 6 | 6 | 6 | 147
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 35 | 37 | 63 | 62 | 66 | 0 | 0 | 0 | 263
    Black or African American | 11 | 11 | 4 | 7 | 4 | 0 | 0 | 0 | 37
    Asian | 0 | 0 | 2 | 2 | 2 | 6 | 6 | 6 | 24
    Other | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Relevant Hypotension up to 6 Hours After the End of Study Drug Infusion
Description: Percentage of participants with clinically relevant hypotension, defined by systolic blood pressure (SBP) < 90 mm Hg (confirmed by a repeated value < 90 mm Hg) or symptoms of hypotension, up to 6 hours after the end of study drug infusion
Time Frame: From start of infusion up to 6 hours post end of infusion
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Percentage of participants
  clinically relevant hypotension | 8.3 [2.32 to 19.98] | 20.4 [10.24 to 34.34] | 18.3 [10.13 to 29.27] | 21.1 [12.33 to 32.44] | 34.7 [23.88 to 46.86] | 0 [0.00 to 45.93] | 33.3 [4.33 to 77.72] | 50.0 [11.81 to 88.19]
  symptoms of hypotension | 2.1 [0.05 to 11.07] | 6.1 [1.28 to 16.87] | 1.4 [0.04 to 7.60] | 2.8 [0.34 to 9.81] | 8.3 [3.12 to 17.26] | 0 [0.00 to 45.93] | 0 [0.00 to 45.93] | 0 [0.00 to 45.93]
  confirmed SBP < 90 mmHg | 6.3 [1.31 to 17.20] | 20.4 [10.24 to 34.34] | 18.3 [10.13 to 29.27] | 21.1 [12.33 to 32.44] | 29.2 [19.05 to 41.07] | 0 [0.00 to 45.93] | 33.3 [4.33 to 77.72] | 50.0 [11.81 to 88.19]
Statistical Analysis 1: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, clinically relevant hypotension - relative risk; Relative risk from placebo = 2.45, 95% CI 2-sided [0.83 to 14.53]
Statistical Analysis 2: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, clinically relevant hypotension - relative difference; Relative difference from placebo = 0.12, 95% CI 2-sided [-0.02 to 0.28]
Statistical Analysis 3: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, symptoms of hypotension - relative risk; Relative risk from placebo = 2.94, 95% CI 2-sided [0.31 to 75.47]
Statistical Analysis 4: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, symptoms of hypotension - relative difference; Relative difference from placebo = 0.04, 95% CI 2-sided [-0.06 to 0.15]
Statistical Analysis 5: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, confirmed SBP < 90 mmHg - relative risk; Relative risk from placebo = 3.27, 95% CI 2-sided [1.01 to 14.66]
Statistical Analysis 6: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.14, 95% CI 2-sided [0.00 to 0.29]
Statistical Analysis 7: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), clinically relevant hypotension - relative risk; Relative risk from placebo = 1.15, 95% CI 2-sided [0.58 to 2.43]
Statistical Analysis 8: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), clinically relevant hypotension - relative difference; Relative difference from placebo = 0.03, 95% CI 2-sided [-0.11 to 0.16]
Statistical Analysis 9: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), symptoms of hypotension - relative risk; Relative risk from placebo = 2.00, 95% CI 2-sided [0.18 to 54.35]
Statistical Analysis 10: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), symptoms of hypotension - relative difference; Relative difference from placebo = 0.01, 95% CI 2-sided [-0.05 to 0.09]
Statistical Analysis 11: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), confirmed SBP < 90 mmHg - relative risk; Relative risk from placebo = 1.15, 95% CI 2-sided [0.58 to 2.43]
Statistical Analysis 12: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.03, 95% CI 2-sided [-0.11 to 0.16]
Statistical Analysis 13: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), clinically relevant hypotension - relative risk; Relative risk from placebo = 1.90, 95% CI 2-sided [1.04 to 3.59]
Statistical Analysis 14: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), clinically relevant hypotension - relative difference; Relative difference from placebo = 0.16, 95% CI 2-sided [0.01 to 0.31]
Statistical Analysis 15: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), symptoms of hypotension - relative risk; Relative risk from placebo = 5.92, 95% CI 2-sided [0.91 to 149.72]
Statistical Analysis 16: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), symptoms of hypotension - relative difference; Relative difference from placebo = 0.07, 95% CI 2-sided [-0.01 to 0.16]
Statistical Analysis 17: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), confirmed SBP < 90 mmHg - relative risk; Relative risk from placebo = 1.59, 95% CI 2-sided [0.87 to 3.21]
Statistical Analysis 18: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.11, 95% CI 2-sided [-0.04 to 0.25]
Statistical Analysis 19: Comparison: Placebo - Part II (Japan Cohort) vs BMS-986231 6 µg/kg/Min - Part II (Japan Cohort); Test type: Superiority — Part II-Japan (low dose), clinically relevant hypotension - relative difference; Relative difference from placebo = 0.33, 95% CI 2-sided [-0.17 to 0.78]
Statistical Analysis 20: Comparison: Placebo - Part II (Japan Cohort) vs BMS-986231 6 µg/kg/Min - Part II (Japan Cohort); Test type: Superiority — Part II-Japan (low dose), confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.33, 95% CI 2-sided [-0.17 to 0.78]
Statistical Analysis 21: Comparison: Placebo - Part II (Japan Cohort) vs BMS-986231 12 µg/kg/Min - Part II (Japan Cohort); Test type: Superiority — Part II-Japan (high dose), clinically relevant hypotension - relative difference; Relative difference from placebo = 0.50, 95% CI 2-sided [-0.04 to 0.88]
Statistical Analysis 22: Comparison: Placebo - Part II (Japan Cohort) vs BMS-986231 12 µg/kg/Min - Part II (Japan Cohort); Test type: Superiority — Part II-Japan (high dose), confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.50, 95% CI 2-sided [-0.04 to 0.88]

2. Secondary Outcome: Change in NT-proBNP From Baseline to Hour 24, 48, 72, 120 or Discharge (Whichever Comes First), and at Day 32
Description: Assess the effect of BMS-986231 on NT-proBNP (N-terminal prohormone of brain natriuretic peptide)
Time Frame: 0, 24, 48, 72, 120 hour or discharge; Day 32
Population: All treated participants
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
pmol/L
  24 hour: number analyzed (Participants) | 43 | 45 | 71 | 71 | 72 | 6 | 6 | 6
  24 hour | -270.88 (400.320) | -364.46 (456.158) | -147.96 (452.239) | -340.74 (430.639) | -416.91 (503.825) | -129.70 (255.716) | -165.93 (185.910) | -397.60 (330.721)
  48 hour: number analyzed (Participants) | 43 | 43 | 71 | 71 | 72 | 6 | 6 | 6
  48 hour | -405.06 (591.711) | -510.51 (592.734) | -210.87 (580.487) | -300.87 (725.268) | -472.32 (610.590) | -329.24 (646.985) | -251.73 (243.794) | -497.35 (725.286)
  72 hour: number analyzed (Participants) | 40 | 38 | 71 | 71 | 72 | 6 | 6 | 6
  72 hour | -396.21 (675.761) | -373.86 (702.530) | -249.26 (655.999) | -118.86 (900.798) | -293.94 (685.681) | -433.08 (761.573) | 9.89 (523.754) | -229.56 (809.850)
  120 hour: number analyzed (Participants) | 29 | 23 | 71 | 71 | 72 | 6 | 6 | 6
  120 hour | -541.36 (773.006) | -409.53 (751.624) | -140.60 (1358.127) | -76.20 (993.110) | -390.21 (717.114) | -434.36 (659.528) | -379.06 (244.917) | -552.55 (824.009)
  Day 32: number analyzed (Participants) | 40 | 42 | 71 | 71 | 72 | 6 | 6 | 6
  Day 32 | -202.07 (799.169) | -91.61 (2254.397) | -321.73 (600.297) | -361.73 (782.881) | -476.86 (716.072) | -556.69 (1288.342) | -343.64 (377.590) | -706.11 (1111.877)

3. Secondary Outcome: Change in Participant-reported Resting Dyspnea From Baseline Through Hour 72
Description: Endpoint was measured by the area under the curve (AUC) of the 11-point Numerical Rating Scale (NRS) obtained at baseline, and Hours 6, 12, 24, 48, and 72.
  Participants were asked to report their absolute current severity of dyspnea on an 11-point numerical rating scale (NRS; range 0 to 10).
  The numerical rating scale (NRS) was used to assess the degree of dyspnea (breathlessness), measured using an 11-point scale provided by the Sponsor.
  A score of 0 represents "I am not breathless at all" and 10 represents "I am the most breathless I can possibly imagine".
Time Frame: Hours 6, 12, 24, 48, and 72
Population: All treated participants
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Scores on a scale
  6 hour: number analyzed (Participants) | 43 | 44 | 68 | 66 | 68 | 6 | 6 | 6
  6 hour | -1.5 (1.84) | -1.5 (1.64) | -1.1 (1.90) | -1.7 (1.94) | -1.7 (2.13) | -0.3 (1.03) | 0.0 (2.90) | -1.3 (3.44)
  12 hour: number analyzed (Participants) | 42 | 42 | 65 | 64 | 66 | 6 | 6 | 6
  12 hour | -2.1 (2.38) | -2.2 (1.73) | -1.7 (2.75) | -2.4 (2.38) | -2.0 (2.49) | -1.0 (1.79) | -0.2 (3.37) | -1.4 (4.22)
  24 hour: number analyzed (Participants) | 44 | 46 | 67 | 67 | 70 | 6 | 6 | 6
  24 hour | -2.0 (2.50) | -2.1 (2.19) | -2.1 (2.82) | -2.9 (2.68) | -2.2 (2.42) | -0.8 (1.72) | -1.5 (3.02) | -1.2 (2.14)
  48 hour: number analyzed (Participants) | 42 | 46 | 66 | 67 | 68 | 6 | 6 | 6
  48 hour | -2.8 (2.15) | -2.6 (2.51) | -2.8 (3.00) | -3.4 (2.44) | -2.8 (2.45) | -1.2 (1.47) | -0.8 (3.43) | -2.0 (1.67)
  72 hour: number analyzed (Participants) | 39 | 39 | 63 | 60 | 68 | 6 | 6 | 6
  72 hour | -2.9 (2.23) | -3.7 (2.22) | -3.2 (3.19) | -3.9 (2.28) | -3.2 (2.73) | -1.2 (2.14) | -1.2 (3.19) | -2.0 (2.00)

4. Secondary Outcome: Percentage of Participants With Symptomatic Hypotension up to 6 Hours After the End of Study Drug Infusion
Description: The percentage of participants experiencing symptoms of hypotension up to 6 hours post-treatment was reported for each arm.
Time Frame: From start of infusion up to 6 hours post end of infusion
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Percentage of participants | 2.1 [0.05 to 11.07] | 6.1 [1.28 to 16.87] | 1.4 [0.04 to 7.60] | 2.8 [0.34 to 9.81] | 8.3 [3.12 to 17.26] | 0 [0.00 to 45.93] | 0 [0.00 to 45.93] | 0 [0.00 to 45.93]
Statistical Analysis 1: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, symptoms of hypotension - relative risk; Relative risk from placebo = 2.94, 95% CI 2-sided [0.31 to 75.47]
Statistical Analysis 2: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, symptoms of hypotension - relative difference; Relative difference from placebo = 0.04, 95% CI 2-sided [-0.06 to 0.15]
Statistical Analysis 3: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), symptoms of hypotension - relative risk; Relative risk from placebo = 2.00, 95% CI 2-sided [0.18 to 54.35]
Statistical Analysis 4: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), symptoms of hypotension - relative difference; Relative difference from placebo = 0.01, 95% CI 2-sided [-0.05 to 0.09]
Statistical Analysis 5: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), symptoms of hypotension - relative risk; Relative risk from placebo = 5.92, 95% CI 2-sided [0.91 to 149.72]
Statistical Analysis 6: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), symptoms of hypotension - relative difference; Relative difference from placebo = 0.07, 95% CI 2-sided [-0.01 to 0.16]

5. Secondary Outcome: Percentage of Participants With SBP < 90 mm Hg (Confirmed by a Repeated Value)
Description: The percentage of participants experiencing SBP < 90 mm Hg (confirmed by a repeated value) up to 6 hours post-treatment was reported for each arm.
Time Frame: From start of infusion up to 6 hours post end of infusion
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Percentage of participants | 6.3 [1.31 to 17.20] | 20.4 [10.24 to 34.34] | 18.3 [10.13 to 29.27] | 21.1 [12.33 to 32.44] | 29.2 [19.05 to 41.07] | 0 [0.00 to 45.93] | 33.3 [4.33 to 77.72] | 50.0 [11.81 to 88.19]
Statistical Analysis 1: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, confirmed SBP < 90 mmHg - relative risk; Relative risk from placebo = 3.27, 95% CI 2-sided [1.01 to 14.66]
Statistical Analysis 2: Comparison: Placebo - Part I vs BMS-986231 - Part I; Test type: Superiority — Part I, confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.14, 95% CI 2-sided [0.00 to 0.29]
Statistical Analysis 3: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), confirmed SBP < 90 mmHg - relative risk; Relative risk from placebo = 1.15, 95% CI 2-sided [0.58 to 2.43]
Statistical Analysis 4: Comparison: Placebo - Part II vs BMS-986231 6 µg/kg/Min - Part II; Test type: Superiority — Part II (low dose), confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.03, 95% CI 2-sided [-0.11 to 0.16]
Statistical Analysis 5: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), confirmed SBP < 90 mmHg - relative risk; Relative risk from placebo = 1.59, 95% CI 2-sided [0.87 to 3.21]
Statistical Analysis 6: Comparison: Placebo - Part II vs BMS-986231 12 µg/kg/Min - Part II; Test type: Superiority — Part II (high dose), confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.11, 95% CI 2-sided [-0.04 to 0.25]
Statistical Analysis 7: Comparison: Placebo - Part II (Japan Cohort) vs BMS-986231 6 µg/kg/Min - Part II (Japan Cohort); Test type: Superiority — Part II-Japan (low dose), confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.33, 95% CI 2-sided [-0.17 to 0.78]
Statistical Analysis 8: Comparison: Placebo - Part II (Japan Cohort) vs BMS-986231 12 µg/kg/Min - Part II (Japan Cohort); Test type: Superiority — Part II-Japan (high dose), confirmed SBP < 90 mmHg - relative difference; Relative difference from placebo = 0.50, 95% CI 2-sided [-0.04 to 0.88]

6. Secondary Outcome: Number of Participants With a Serious Adverse Events (SAE) Assessed up to Day 32
Description: Number of participants who experienced an in-study SAE.
  Medical Dictionary for Regulatory Activities (MedDRA) version: 22.0 Included serious adverse events with onset time from the start of study treatment, up to and including 32 days after the start of study treatment.
Time Frame: 32 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Participants | 11 | 14 | 23 | 15 | 15 | 1 | 0 | 1

7. Secondary Outcome: Number of Participants Who Discontinued Due to Hypotension
Description: Number of participants who discontinued study treatment due to hypotension.
  Medical Dictionary for Regulatory Activities (MedDRA) version: 22.0
  Included nonserious adverse events with onset time from the start of study treatment, up to and including 120 hours after the start of study treatment and serious adverse events with onset time from the start of study treatment, up to and including 32 days after the start of study treatment.
  Hypotension defined as systolic blood pressure (SBP) < 90 mmHg.
Time Frame: up to 120 hours (for AEs); up to 32 days (for SAEs)
Population: All treated participants
  Note: Discontinuation due to hypotension occurred per protocol-mandated lowering of blood pressure to < 90 mmHg.
Measure: Number; unit: Participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Participants | 4 | 8 | 7 | 13 | 16 | 0 | 1 | 3

8. Secondary Outcome: Number of Participants Who Discontinued, Experienced a Down-titration or Dose Interruption Due to Decreased Blood Pressure
Description: Number of participants who discontinued study treatment, experienced a down-titration (dose reduction) or dose interruption due to decreased blood pressure/hypotension are reported below.
  Medical Dictionary for Regulatory Activities (MedDRA) version: 22.0
  Included nonserious adverse events with onset time from the start of study treatment, up to and including 120 hours after the start of study treatment and serious adverse events with onset time from the start of study treatment, up to and including 32 days after the start of study treatment.
  If the participant experienced systolic blood pressure (SBP) < 95 mm Hg, without symptoms related to hypotension, the measurement was repeated within 15 minutes. If the SBP remained < 95 mm Hg, the dose reduction occurred.
Time Frame: up to 120 hours (for AEs); up to 32 days (for SAEs)
Population: All treated participants
  Note: Discontinuation due to decreased blood pressure occurred per protocol-mandated lowering of blood pressure to < 95 mmHg.
Measure: Number; unit: Participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Participants
  discontinuation | 4 | 8 | 7 | 13 | 15 | 0 | 1 | 3
  down-titration | 3 | 9 | 9 | 10 | 25 | 0 | 1 | 3
  interruption | 3 | 4 | 4 | 12 | 13 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With an Adverse Event (AE) Assessed up to 120 Hours
Description: Number of participants who experienced an in-study AE.
  Medical Dictionary for Regulatory Activities (MedDRA) version: 22.0
  Included nonserious adverse events with onset time from the start of study treatment, up to and including 120 hours after the start of study treatment.
Time Frame: up to 120 hours
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Participants | 31 | 39 | 48 | 48 | 55 | 2 | 6 | 6

10. Secondary Outcome: Number of Participants Who Died (All- Cause and Cardiovascular-related) Through Day 182
Description: Number of participants who died (all- cause and CV related) through Day 182.
  Medical Dictionary for Regulatory Activities (MedDRA) version: 22.0
  CV=Cardiovascular
Time Frame: through 182 days
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Participants
  All-cause | 3 [1.31 to 17.20] | 3 [1.28 to 16.87] | 11 [8.00 to 26.03] | 12 [9.05 to 27.66] | 9 [5.88 to 22.41] | 0 [0.00 to 45.93] | 0 [0.00 to 45.93] | 1 [0.42 to 64.12]
  CV-related | 3 [1.31 to 17.20] | 2 [0.50 to 13.98] | 9 [5.96 to 22.70] | 10 [6.97 to 24.38] | 4 [1.53 to 13.62] | 0 [0.00 to 45.93] | 0 [0.00 to 45.93] | 0 [0.00 to 45.93]

11. Secondary Outcome: Change in Troponin T From Baseline to Hour 24, 48, and 72
Description: Baseline = Last non-missing result with a collection date-time less than or on the date-time of the start of infusion of study drug
Time Frame: from baseline to Hour 24, 48, and 72
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
ng/L
  24 hour: number analyzed (Participants) | 41 | 44 | 69 | 66 | 68 | 6 | 6 | 6
  24 hour | 4.11 (27.303) | -1.31 (12.278) | -1.80 (11.266) | -3.45 (20.030) | -8.09 (37.864) | -4.67 (3.983) | 1.33 (5.750) | -7.67 (16.669)
  48 hour: number analyzed (Participants) | 41 | 44 | 64 | 63 | 68 | 6 | 6 | 6
  48 hour | -0.93 (22.714) | 14.56 (81.979) | -2.88 (16.424) | 8.08 (71.672) | -11.15 (45.495) | -10.67 (10.633) | 49.50 (118.417) | -8.40 (25.501)
  72 hour: number analyzed (Participants) | 39 | 38 | 63 | 57 | 65 | 6 | 6 | 6
  72 hour | 6.07 (30.033) | 6.76 (66.673) | -1.44 (16.472) | 5.00 (65.766) | -13.05 (68.276) | -10.50 (12.145) | 248.00 (433.581) | -15.00 (25.169)

12. Secondary Outcome: Number of Participants With Marked Laboratory Abnormality Assessed to 120 Hours - Hematology
Description: Number of participants who experienced an in-study Hematology marked laboratory abnormality (reported in > 5% of total participants).
  Medical Dictionary for Regulatory Activities (MedDRA) version: 22.0
Time Frame: to 120 hours
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Participants
  high leukocyte counts: number analyzed (Participants) | 47 | 49 | 71 | 68 | 72 | 6 | 6 | 6
  high leukocyte counts | 5 | 2 | 5 | 4 | 3 | 0 | 0 | 0
  low hemoglobin values: number analyzed (Participants) | 47 | 49 | 71 | 68 | 72 | 6 | 6 | 6
  low hemoglobin values | 4 | 5 | 5 | 6 | 4 | 1 | 1 | 0
  low platelet values: number analyzed (Participants) | 47 | 49 | 71 | 67 | 72 | 6 | 6 | 6
  low platelet values | 4 | 2 | 2 | 7 | 1 | 0 | 0 | 0
  low neutrophils values: number analyzed (Participants) | 46 | 49 | 71 | 67 | 72 | 6 | 6 | 6
  low neutrophils values | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  low leukocyte counts: number analyzed (Participants) | 48 | 49 | 71 | 68 | 72 | 6 | 6 | 6
  low leukocyte counts | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  low hematocrit values: number analyzed (Participants) | 48 | 49 | 71 | 68 | 72 | 6 | 6 | 6
  low hematocrit values | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0
  low erythrocytes values: number analyzed (Participants) | 48 | 49 | 71 | 68 | 72 | 6 | 6 | 6
  low erythrocytes values | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Marked Laboratory Abnormality Assessed to 120 Hours - Chemistry
Description: Number of participants who experienced an in-study Chemistry marked laboratory abnormality (reported in > 5% of total participants).
  Medical Dictionary for Regulatory Activities (MedDRA) version: 22.0
Time Frame: to 120 hours
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Participants
  high blood urea nitrogen values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high blood urea nitrogen values | 23 | 16 | 23 | 23 | 18 | 0 | 1 | 2
  high urate values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high urate values | 10 | 15 | 10 | 20 | 8 | 0 | 1 | 1
  high potassium values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high potassium values | 2 | 5 | 6 | 7 | 2 | 0 | 1 | 0
  high alanine aminotransferase (ALT) values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high alanine aminotransferase (ALT) values | 6 | 1 | 5 | 2 | 2 | 0 | 0 | 0
  high alkaline phosphatase values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high alkaline phosphatase values | 5 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  low protein values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  low protein values | 3 | 9 | 3 | 8 | 4 | 0 | 1 | 0
  high asparate aminotransferase values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high asparate aminotransferase values | 4 | 0 | 4 | 2 | 1 | 0 | 0 | 0
  high bilirubin values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high bilirubin values | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0
  high bicarbonate values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high bicarbonate values | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  low chloride counts: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  low chloride counts | 1 | 2 | 1 | 4 | 1 | 0 | 0 | 0
  high creatine kinase values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high creatine kinase values | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  high protein values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high protein values | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
  high sodium values: number analyzed (Participants) | 47 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  high sodium values | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  low bicarbonate values: number analyzed (Participants) | 48 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  low bicarbonate values | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
  low sodium values: number analyzed (Participants) | 48 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  low sodium values | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  low albumin values: number analyzed (Participants) | 48 | 49 | 71 | 69 | 72 | 6 | 6 | 6
  low albumin values | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  low calcium values: number analyzed (Participants) | 48 | 49 | 71 | 68 | 72 | 6 | 6 | 6
  low calcium values | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Marked Laboratory Abnormality Assessed to 120 Hours - Urinalysis
Description: Number of participants who experienced an in-study Urinalysis marked laboratory abnormality (reported in > 5% of total participants).
  Medical Dictionary for Regulatory Activities (MedDRA) version: 22.0
Time Frame: to 120 hours
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
Participants
  high protein values: number analyzed (Participants) | 45 | 48 | 61 | 64 | 69 | 6 | 6 | 5
  high protein values | 10 | 11 | 16 | 13 | 17 | 2 | 2 | 2
  high erythrocyte values: number analyzed (Participants) | 28 | 38 | 47 | 47 | 50 | 5 | 5 | 4
  high erythrocyte values | 1 | 1 | 1 | 3 | 2 | 0 | 0 | 0
  high leukocytes values: number analyzed (Participants) | 48 | 49 | 47 | 47 | 50 | 5 | 5 | 4
  high leukocytes values | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0

15. Secondary Outcome: Change in Vital Signs From Baseline to 120 Hours - Blood Pressure
Description: The change in baseline for vital signs was reported for each arm.
Time Frame: to 120 hours
Population: All treated participants with a 120-hour evaluation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 29 | 26 | 50 | 48 | 44 | 6 | 6 | 6
mmHg
  systolic blood pressure, mmHg | -6.8 (16.60) | 0.0 (17.75) | -4.3 (15.23) | -7.9 (15.60) | -8.8 (14.01) | -10.3 (15.60) | -17.5 (9.14) | -6.2 (16.44)
  diastolic blood pressure, mmHg | -4.0 (12.67) | -1.9 (13.53) | -4.4 (12.99) | -3.4 (14.37) | -1.6 (10.83) | 1.7 (16.24) | -15.7 (19.08) | -9.3 (14.45)

16. Secondary Outcome: Change in Vital Signs From Baseline to 120 Hours - Heart Rate
Description: The change in baseline for vital signs was reported for each arm.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
beats/min | -1.8 (15.53) | -9.1 (17.13) | -8.3 (15.55) | -4.6 (15.40) | -6.3 (15.60) | -6.7 (21.88) | -3.0 (13.31) | 3.8 (11.55)

17. Secondary Outcome: Change in Vital Signs From Baseline to 120 Hours - Respiratory Rate
Description: The change in baseline for vital signs was reported for each arm.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
breaths/min | -2.6 (3.93) | -3.0 (4.82) | -2.9 (3.80) | -2.6 (4.33) | -1.8 (3.96) | -2.3 (2.88) | 0.0 (9.98) | -1.4 (3.58)

18. Secondary Outcome: Change in Vital Signs From Baseline to 120 Hours - Temperature
Description: The change in baseline for vital signs was reported for each arm.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
degrees C | -0.04 (0.643) | 0.09 (0.649) | 0.04 (0.427) | 0.00 (0.342) | -0.05 (0.481) | -0.47 (0.650) | -0.27 (0.535) | 0.44 (0.541)

19. Secondary Outcome: Change in Electrocardiograms (ECGs) From Baseline to 120 Hours - Mean Heart Rate
Description: The change in baseline for ECGs was reported for each arm.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 5 | 6 | 6
beats/min | -5.3 (9.36) | -6.8 (21.31) | -7.1 (17.46) | -5.1 (18.64) | -6.1 (17.33) | 2.0 (10.72) | -13.0 (12.62) | -5.2 (14.85)

20. Secondary Outcome: Change in Electrocardiograms (ECGs) From Baseline to 120 Hours - PR, QT, QTcF Intervals and QRS Duration
Description: The change in baseline for ECGs was reported for each arm.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
msec
  PR Interval, Aggregate, msec: number analyzed (Participants) | 17 | 12 | 19 | 26 | 23 | 4 | 5 | 4
  PR Interval, Aggregate, msec | -17.4 (66.31) | -2.3 (32.11) | -0.1 (23.49) | 10.9 (22.02) | 2.0 (25.41) | -1.5 (16.50) | 10.4 (26.32) | 6.0 (30.10)
  QRS Duration, Aggregate, msec: number analyzed (Participants) | 26 | 21 | 43 | 43 | 44 | 5 | 6 | 6
  QRS Duration, Aggregate, msec | 5.1 (22.19) | -0.1 (12.46) | 1.6 (20.29) | -1.6 (13.22) | 2.7 (16.77) | -3.0 (4.80) | -2.5 (7.20) | 3.0 (4.38)
  QT Interval, Aggregate, msec: number analyzed (Participants) | 25 | 20 | 41 | 42 | 44 | 5 | 6 | 6
  QT Interval, Aggregate, msec | -10.6 (49.20) | 7.2 (48.25) | 8.7 (53.17) | 5.8 (42.19) | -0.3 (45.39) | -30.0 (28.17) | 5.7 (24.41) | 16.5 (50.22)
  QTcF Interval, Aggregate, msec: number analyzed (Participants) | 25 | 21 | 41 | 43 | 44 | 5 | 6 | 6
  QTcF Interval, Aggregate, msec | -27.5 (41.79) | -13.9 (41.56) | -4.0 (51.04) | -4.0 (33.59) | -10.3 (37.63) | -24.8 (20.00) | -8.8 (22.35) | 3.2 (22.93)

21. Secondary Outcome: Change in Physical Measurements From Baseline to 120 Hours
Description: The change in baseline for physical measurements was reported for each arm.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72 | 6 | 6 | 6
kg | 0.00 (0383) | 0.10 (0.285) | -2.87 (4.447) | -2.96 (4.231) | -1.83 (5.295) | -3.58 (2.182) | -3.97 (2.160) | -6.08 (4.009)

22. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Main Study Cohorts Only - x10^9 Cells/L
Description: The change in baseline for laboratory assessments was reported for each arm of the Main study cohorts only.
Time Frame: to 120 hours
Population: All treated participants with a 120-hour evaluation
Measure: Mean (Standard Deviation); unit: x10^9 cells/L
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II
Number analyzed (Participants) | 30 | 23 | 41 | 36 | 39
x10^9 cells/L
  leukocyte, x10^9 c/L | 0.12 (3.078) | -1.38 (1.892) | -0.20 (4.370) | 0.20 (2.549) | -0.09 (1.980)
  platelet, x10^9 c/L: number analyzed (Participants) | 30 | 22 | 38 | 34 | 38
  platelet, x10^9 c/L | 5.63 (31.679) | -5.77 (34.666) | 1.84 (40.808) | 3.26 (37.888) | 1.26 (31.135)

23. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Main Study Cohorts Only - g/L
Description: The change in baseline for laboratory assessments was reported for each arm of the Main study cohorts only.
Time Frame: to 120 hours
Population: All treated participants with a 120-hour evaluation
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II
Number analyzed (Participants) | 30 | 23 | 46 | 42 | 43
g/L
  hemoglobin, g/L: number analyzed (Participants) | 30 | 23 | 41 | 36 | 39
  hemoglobin, g/L | -0.67 (11.851) | -0.70 (8.573) | 1.20 (11.487) | 0.94 (11.684) | 1.38 (9.161)
  protein, g/L: number analyzed (Participants) | 30 | 22 | 46 | 42 | 43
  protein, g/L | 1.10 (6.172) | 2.77 (5.839) | 0.57 (8.178) | 0.38 (6.048) | -0.05 (5.367)

24. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Main Study Cohorts Only - mmol/L
Description: The change in baseline for laboratory assessments was reported for each arm of the Main study cohorts only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72
mmol/L
  blood urea nitrogen, mmol/L: number analyzed (Participants) | 30 | 23 | 48 | 45 | 46
  blood urea nitrogen, mmol/L | 4.01 (5.474) | 0.32 (3.164) | 1.96 (3.920) | 2.15 (5.016) | 1.24 (3.655)
  urate, mmol/L: number analyzed (Participants) | 30 | 22 | 46 | 43 | 42
  urate, mmol/L | 0.06 (0.154) | 0.01 (0.108) | -0.01 (0.126) | 0.04 (0.147) | -0.03 (0.111)
  potassium, mmol/L: number analyzed (Participants) | 30 | 23 | 49 | 46 | 46
  potassium, mmol/L | 0.19 (0.697) | 0.28 (0.513) | 0.21 (0.692) | 0.13 (0.558) | 0.15 (0.651)

25. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Main Study Cohorts Only - U/L
Description: The change in baseline for laboratory assessments was reported for each arm of the Main study cohorts only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72
U/L
  alanine aminotransferase (ALT), U/L: number analyzed (Participants) | 30 | 22 | 46 | 42 | 43
  alanine aminotransferase (ALT), U/L | 148.13 (837.833) | -2.73 (11.089) | -3.22 (102.038) | 30.36 (189.310) | -13.07 (76.357)
  alkaline phosphatase, U/L: number analyzed (Participants) | 30 | 23 | 48 | 44 | 45
  alkaline phosphatase, U/L | -1.00 (28.018) | 1.65 (11.052) | -1.31 (25.186) | 5.43 (26.007) | -0.49 (21.474)
  asparate aminotransferase, U/L: number analyzed (Participants) | 30 | 22 | 46 | 43 | 43
  asparate aminotransferase, U/L | 214.77 (1204.410) | -2.77 (10.277) | -11.15 (127.903) | 10.81 (65.009) | -10.00 (52.075)

26. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Main Study Cohorts Only - mg/dL
Description: The change in baseline for laboratory assessments was reported for each arm of the Main study cohorts only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72
mg/dL | NA (NA) — 120 hour data not collected | NA (NA) — 120 hour data not collected | NA (NA) — 120 hour data not collected | NA (NA) — 120 hour data not collected | NA (NA) — 120 hour data not collected

27. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Main Study Cohorts Only - x10^12 c/L
Description: The change in baseline for laboratory assessments was reported for each arm of the Main study cohorts only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: x10^12 c/L
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II
Number analyzed (Participants) | 48 | 49 | 71 | 71 | 72
x10^12 c/L | -0.02 (0.394) | 0.02 (0.305) | 0.04 (0.409) | 0.04 (0.481) | 0.09 (0.337)

28. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Japan Cohort Only - Protein (Nmol/L)
Description: The change in baseline for laboratory assessments was reported for each arm of the Japan cohort only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 6 | 6 | 5
nmol/L | 79.38 (192.568) | 74.13 (110.919) | 131.64 (407.611)

29. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Japan Cohort Only - Creatinine (µmol/L)
Description: The change in baseline for laboratory assessments was reported for each arm of the Japan cohort only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 6 | 6 | 5
µmol/L | 4.33 (17.728) | -1.50 (6.775) | 12.40 (23.891)

30. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Japan Cohort Only - Cystatin (mg/L)
Description: The change in baseline for laboratory assessments was reported for each arm of the Japan cohort only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 6 | 6 | 5
mg/L | 0.18 (0.268) | 0.17 (0.150) | 0.25 (0.077)

31. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Japan Cohort Only - Percentage Fractional Potassium Excretion
Description: The change in baseline for laboratory assessments was reported for each arm of the Japan cohort only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: Fractional Potassium Excretion percent
Arm/Group | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 6 | 5 | 5
Fractional Potassium Excretion percent | 4.88 (8.009) | -1.22 (4.926) | -12.34 (13.316)

32. Secondary Outcome: Change in Laboratory Assessments From Baseline to 120 Hours, Japan Cohort Only - Percentage Fractional Sodium Excretion
Description: The change in baseline for laboratory assessments was reported for each arm of the Japan cohort only.
Time Frame: to 120 hours
Population: All treated participants
Measure: Mean (Standard Deviation); unit: Fractional Sodium Excretion percent
Arm/Group | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
Number analyzed (Participants) | 6 | 6 | 5
Fractional Sodium Excretion percent | 0.02 (2.076) | -2.62 (4.538) | -5.50 (7.984)

ADVERSE EVENTS:
Time Frame: Includes non-serious adverse events with onset time from the start of study treatment, up to and including 120 hours after the start of study treatment and serious adverse events with onset time from the start of study treatment, up to and including 32 days after the start of study treatment. Mortality data reported through 182 days post-treatment
Arm/Group | Placebo - Part I | BMS-986231 - Part I | Placebo - Part II | BMS-986231 6 µg/kg/Min - Part II | BMS-986231 12 µg/kg/Min - Part II | Placebo - Part II (Japan Cohort) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort)
All-Cause Mortality (participants affected / at risk) | 3/48 | 3/49 | 11/71 | 12/71 | 9/72 | 0/6 | 0/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 11/48 | 14/49 | 23/71 | 15/71 | 15/72 | 1/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 18/48 | 40/49 | 47/71 | 43/71 | 54/72 | 2/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part I (N=48) | BMS-986231 - Part I (N=49) | Placebo - Part II (N=71) | BMS-986231 6 µg/kg/Min - Part II (N=71) | BMS-986231 12 µg/kg/Min - Part II (N=72) | Placebo - Part II (Japan Cohort) (N=6) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) (N=6) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort) (N=6)
CARDIAC FAILURE (Cardiac disorders) | 2 | 6 | 8 | 2 | 7 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
CARDIORENAL SYNDROME (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ACINETOBACTER BACTERAEMIA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ENDOCARDITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
DELIRIUM (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ORGANIC BRAIN SYNDROME (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
BLADDER MASS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
END STAGE RENAL DISEASE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ELECTROCARDIOGRAM QRS COMPLEX PROLONGED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANGIOPATHY (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ILIAC ARTERY OCCLUSION (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
HEPATIC CONGESTION (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part I (N=48) | BMS-986231 - Part I (N=49) | Placebo - Part II (N=71) | BMS-986231 6 µg/kg/Min - Part II (N=71) | BMS-986231 12 µg/kg/Min - Part II (N=72) | Placebo - Part II (Japan Cohort) (N=6) | BMS-986231 6 µg/kg/Min - Part II (Japan Cohort) (N=6) | BMS-986231 12 µg/kg/Min - Part II (Japan Cohort) (N=6)
HYPOTENSION (Vascular disorders) | 5 | 14 | 15 | 20 | 31 | 0 | 3 | 4
CARDIAC FAILURE (Cardiac disorders) | 2 | 6 | 8 | 2 | 7 | 0 | 0 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 6 | 5 | 4 | 2 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 4 | 3 | 1 | 2 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 7 | 8 | 8 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 2 | 2 | 6 | 2 | 1 | 1 | 1 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 3 | 0 | 3 | 2 | 1 | 0 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 2 | 0 | 3 | 3 | 0 | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VITREOUS DETACHMENT (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03016325/SAP_001.pdf
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03016325/Prot_002.pdf